CLINICAL TRIAL: NCT01696409
Title: The Effect of Vitamin D on Measures of Bone Health and Gene Expression
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Michael F. Holick, Dr. Michael Holick, Boston University
Other Study IDs: Vitamin D and Gene Expression
Record Dates: First submitted 2012-06-25; First posted 2012-10-01 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buffy coat has been retained from whole blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm A: 400 IU vitamin D3 once a day for 2 months
  Interventions: Dietary Supplement: 400 IU vitamin D3
- Arm B: 2000 IU Vitamin D3 once/day for 2 months
  Interventions: Dietary Supplement: 2000 IU vitamin D3

INTERVENTIONS:
Dietary Supplement: 400 IU vitamin D3 — Take 400 IU once/day for 2 months
  Groups: Arm A
Dietary Supplement: 2000 IU vitamin D3 — 2000 IU vitamin D3 once/day for 2 months
  Groups: Arm B

SUMMARY:
Vitamin D deficiency is now recognized as one of the most common vitamin deficiencies in adults in the United States. Vitamin D deficiency has been connected to many chronic health diseases. The goal of this innovative research is to identify how vitamin D is able to have such wide ranging health benefits. This study will determine which genes are turned on and turned off in adults who receive 2000 IU vitamin D3 per day compared to 400 IU vitamin D3 per day. Results should provide important new insights about the health benefits of vitamin D for adults.

DETAILED DESCRIPTION:
Vitamin D, commonly known as the sunshine vitamin, is produced in the skin from sun exposure as well as from dietary sources. However, very few foods naturally contain vitamin D and the amount of vitamin D in fortified foods typically, 100 IU per serving, has been totally inadequate in satisfying adults vitamin D requirement, which is now been estimated to be at least 2,000 IU of vitamin D a day. As a result, vitamin D deficiency is rapidly being recognized world-wide as the most common vitamin deficiency. Upwards of 50-100% of children and adults have been reported as being vitamin D deficient depending on ethnicity, latitude and skin pigmentation. The investigators reported in women at the time of delivery that 76% of mothers and 81% of newborns were vitamin D deficient despite the fact that the mother was taking a prenatal vitamin containing 400 IU vitamin D and drinking two glasses of milk a day. The investigators also reported 30-80% vitamin D deficiency rates in white and black children, healthy young, middle aged and older adults. There have been numerous epidemiologic and clinical observations relating vitamin D deficiency to many chronic diseases and there are many isolated but no comprehensive studies evaluating various genes that are either suppressed or enhanced by 1,25-dihydroxyvitamin D [1,25(OH)2D]. It has been estimated that upwards of 2000 genes are directly or indirectly influence by 1,25(OH)2 D. To date, however, there have not been any genomic signatures identified in humans in response to correction of vitamin D deficiency. The goal of this pilot study is to determine whether or not vitamin D3 supplementation will affect biomarkers for calcium and bone metabolism, and how they alter gene expression biomarkers, especially genes related to the non-skeletal actions of vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults of all races ages 18 years and older

Exclusion Criteria:

* 1. Pregnant and lactating women.

  2. Current or recent history of hepatic or renal disease

  3. History of taking a daily supplement that contains more than 400 IU vitamin D2 or vitamin D3 within the past month or taking a pharmacologic amount of vitamin D2 or one of the active vitamin D analogs including Zemplar (Paricalcitol), Dovonex (calcipotriol), Hectorol (vitamin D pro hormone)

  4. Subjects who are taking antiseizure medications or glucocorticoids.

  5. Exposure to a tanning bed or tanning on a beach for more than eight hours within the past month.

  6. Known history of elevated calcium. (> 10.5 mg% (mg/dl))

  7. History of intestinal malabsorption (i.e. Cystic Fibrosis, Fat Malabsorption Syndrome, Crohn's Disease)

  8. Unwilling to consent to this trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Students from Boston University Medical School
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Gene Expression | Baseline and Final Visits
  Measurement of mRNA levels from genes specific to bone, calcium, and non-skeletal functions.

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Holick, PhD, MD, Principal Investigator — BUMC
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hossein-nezhad A, Spira A, Holick MF. Influence of vitamin D status and vitamin D3 supplementation on genome wide expression of white blood cells: a randomized double-blind clinical trial. PLoS One. 2013;8(3):e58725. doi: 10.1371/journal.pone.0058725. Epub 2013 Mar 20. PMID 23527013